CLINICAL TRIAL: NCT01280305
Title: A Randomized Trial Administering Raloxifene vs Placebo as add-on to Antipsychotics in Post Menopausal Patients With Schizophrenia or Schizoaffective Disorder
Brief Title: Raloxifene in Treatment of Schizophrenia and Schizoaffective Disorder
Acronym: RAL-S-01
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Mark Weiser MD, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-10-8287-MW-SHEBA
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- raloxifene (Experimental)
  Interventions: Drug: raloxifene
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: raloxifene — raloxifene 60 mg bid
  Arms: raloxifene
Drug: placebo — Placebo bid
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the efficacy of raloxifene compared to placebo, as add-on to anti-psychotics in the treatment of post menopausal patients with schizophrenia.

DETAILED DESCRIPTION:
Epidemiological evidence shows a potentially protective role for estrogen in women with schizophrenia. The onset of schizophrenia is later in woman than in men, with generally a less severe course until after the menopause, when for many women, reductions in estrogen levels appear to trigger an exacerbation or illness (Hafner 2003). ERα (Estrogen receptor alpha) expression is known to be reduced in schizophrenia (Wong, Woon et al. 2010). Raloxifene is a selective estrogen receptor modulator that acts as an estrogen antagonist in breast tissue and may have agonistic actions in the brain. Several studies (Kulkarni, Riedel et al. 2001; Chua, de Izquierdo et al. 2005; Kulkarni, Gurvich et al. 2010) indicate that treatment with estrogen and raloxifene improves symptoms in females with schizophrenia, and recently they showed an improvement in PANSS score in post menopausal women with schizophrenia receiving 60-120mg/d of raloxifene compared to placebo

ELIGIBILITY:
Inclusion Criteria:

1. Post menopausal females: Post menopausal defined as: Women 45 years of age and older with no vaginal bleeding for at least 2 years prior to randomization, and both serum estradiol <73 pmol/L (20 pg/mL) and FSH >30 IU/L (30 mIU/mL).
2. 45-65 years old
3. Willing and able to provide informed consent, after the nature of the study has been fully explained.
4. Current DSM-IV-TR diagnosis of schizophrenia or schizoaffective disorder as confirmed by modified SCID and having had at least 2 prior schizophrenic episodes, or continually ill for at least 6 months.
5. Symptoms: 4 (moderate) or above on CGI-S and 4 (moderate) score or above on two of the following four PANSS items: delusions, hallucinatory behaviors, conceptual disorganization or suspiciousness/ persecution, and/or a total PANSS negative symptoms score of 18.
6. Must be on any antipsychotic drug, for at least 2 weeks prior to the baseline visit, at doses within the PORT criteria, whenever possible. Patients receiving higher doses will have their records reviewed to insure that the dose is required and, if possible, will be stabilized on a lower dose prior to study entry.
7. Inpatients or outpatients. Inpatients will be randomized 3 days or more after admission.

Exclusion Criteria:

1. Unwilling or unable, in the opinion of the Investigator, to comply with study instructions
2. Women of child bearing potential.
3. Women who have amenorrhea due to causes other than natural or surgical menopause i.e. eating disorders or exercise
4. Unstable medical disease (malignancy, poorly controlled diabetes, active ischemic cardiac disease, or cardiomyopathy, serious pulmonary disease, kidney disease, impaired liver functioning.
5. Patients treated with cholestyramine, warfarin or concurrent systemic estrogen therapy
6. Likely allergy or sensitivity to raloxifene.
7. At significant risk of committing suicide, or in the opinion of the Investigator, currently is at imminent risk of suicide or harming others.
8. Patients with a current DSM-IV substance or alcohol abuse. Patients with a history of and/or current recreational use of cannabinoids or alcohol, and/or patients who smoke cigarettes can be included.
9. Concurrent delirium, mental retardation, drug-induced psychosis, or history of brain trauma.
10. Patients with hypercoaguable conditions or risk of venous thrombosis.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
PANSS total score at the end of the trial. | 3 times
  PANSS will be assesed at weeks 5, 8 and end of study.

SECONDARY OUTCOMES:
PANSS,CGI-S, CGI-I, BACS and rates of drop outs before the end of the trial. | PANSS 3 times, CGI-S and CGI-I 5 times and BACS 2 times
  PANSS will be assessed at week 5, 8, and end of study; CGI-S, CGI-I, will be assessed at week 2, 5, 8, 12, and end of study; BACS will be assessed at week 8 and end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Weiser, MD, Principal Investigator — Sheba Medical Center
Locations (7):
- Sheba Medical Center, Ramat Gan, Israel
- Romania (6):
  - Clinica de Psihiatrie, Arad, Arad
  - Spitalul de Psihiatrie Botosani, Botoșani
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Alex. Obregia", Bucharest
  - Sp. Jud. "Prof. Dr.O. Fodor", Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Cluj, Cluj-Napoca
  - Spitalul Clinic de Psihiatrie Socola, Iasi, Iași

REFERENCES:
- [Derived] Weiser M, Levi L, Burshtein S, Hagin M, Matei VP, Podea D, Miclutia I, Tiugan A, Pacala B, Grecu IG, Noy A, Zamora D, Davis JM. Raloxifene Plus Antipsychotics Versus Placebo Plus Antipsychotics in Severely Ill Decompensated Postmenopausal Women With Schizophrenia or Schizoaffective Disorder: A Randomized Controlled Trial. J Clin Psychiatry. 2017 Jul;78(7):e758-e765. doi: 10.4088/JCP.15m10498. PMID 28541645